CLINICAL TRIAL: NCT01231165
Title: Comparative Randomized Single-blind Trial of Amiloride in Coronary Heart Disease
Brief Title: Treatment of Coronary Heart Disease With Amiloride
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Carabobo (Other)
Collaborators: Clinical Research Unit at the Docent Institute of Urology (Unknown); Northern Metropolitan Hospital (Unknown); Venezuelan Foundation of Heart Failure (Other)
Responsible Party: Principal Investigator, Antonio Delgado Leon, MD, Prof. of Medicine, MD, University of Carabobo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UIC-5 2008
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Amiloride; Nitrates; WW Domain-Containing Oxidoreductase; Clopidogrel; Aspirin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amiloride,nitrates,clopidogrel,aspirin,statins (Experimental): Comparative Efficacious Research
  Interventions: Drug: Amiloride
- Nitrates, clopidogrel, aspirin, statins (Active Comparator): Comparative Efficacious Research
  Interventions: Drug: Nitrates, clopidogrel, aspirin, statins

INTERVENTIONS:
Drug: Amiloride — 5mg/daily for 12th months
  Other Names: Nitrates (40mg/daily) for 12 months; Clopidogrel(75mg/daily)for 12 months; Aspirin (80mg/daily) for 12 months; Statins (20mg/daily) for 12 months
  Arms: Amiloride,nitrates,clopidogrel,aspirin,statins
Drug: Nitrates, clopidogrel, aspirin, statins — Comparative Efficacious Research
  Other Names: Nitrates (40mg/daily) for 12 months; Clopidogrel(75mg/daily)for 12 months; Aspirin (80mg/daily) for 12 months; Statins (20mg/daily) for 12 months
  Arms: Nitrates, clopidogrel, aspirin, statins

SUMMARY:
Treatment of coronary artery disease is a major health care problem across the entire word, and the United States. Unfortunately, despite a number of medical advances, diagnostic procedure, or epidemiological studies, the treatment of these patients remain complex, and and at times frustrating. In fact, the COURAGE trial conducted in 50 centers across United States and Canada documented that drug treatment, coronary interventions or both were not effective solution in coronary artery diseases.

A novel approach has recently been developed, based on the critical role of the potassium (K) content in red-blood-cell in myocardial oxygenation, since oxygen and K binding by hemoglobin (red-blood-cell) occurs simultaneously in blood passing through the lungs, whereas in the organs as the heart, the hemoglobin release both Oxygen and K ions.

This apparently simple mechanisms occurs in human blood in all individuals but could be altered in subjects with acquired or hereditable defect in red-blood-cell K content. The purpose of this trial, thus, will be to evaluate the pharmacological effects of Amiloride on RBC K-uptake and transport and its impact on reversion of angina, electrocardiographic changes of myocardial ischemia and electrical regeneration of the heart in subjects with coronary artery diseases.

DETAILED DESCRIPTION:
The Problem: Treatment of Cardiovascular Diseases (CVD) is a major health care problem across the entire word, and particularly in the United States, Japan and European Countries (1). In fact, these life-threatening disorders are a major cause of emergency medical care and hospitalization in the United States, and according the National Center for Health Statistics (NCHS) there were approximately 1,565,000 hospitalizations for primary or secondary diagnosis of an acute coronary syndrome (ACS), 669,000 for unstable angina (UA) and 896,000 for myocardial infarction (MI). In the 2003, NCHS reported 4,497,000 visits to emergency departments for primary diagnosis of CVD, wherein the average age of a person having a first heart attack is calculated at 65.8 years for men and 70.4 years for women (2)

Although the treatment of angina, chest pain secondary to coronary heart disease (stable chronic angina) and one of the most common and early symptom of Coronary Heart Disease (CHD) can be tracked as far as 1880's, it still represents a medically unresolved problem. Indeed, treatment of angina in particular, as well as associated condition as ACS, UA, and MI, involves a large number of life-style recommendations, dietetic advice, drugs, coronary artery intervention, or coronary bypass surgery aimed to improve symptoms, quality of life of patients, and even primary or secondary prevention of the stable chronic angina. Unfortunately, despite a century of medical advances and epidemiological studies, the current approach to CVD and coronary heart disease remain complex, and at times frustrating.

Among the proposals to treat stable chronic angina new aspects have been considered, including the single "polypill" agent (aspirin + statin + 3 blood pressure lowering agents in half dose, and folic acid), Simvastatin and intravascular ultrasound study, or intra-coronary angiogenesis therapy (3-5). However, most of them are unpractical, whereas it is difficult to determine whether these changes will translate to meaningful reductions in clinical events, or whether results in highly selected patient populations can be matched to the real-world of prevention and treatment of coronary artery syndromes.

Further, a recent large clinical trial, COURAGE study (6), conducted in 50 hospital centers in the United States and Canada showed that optimal drug treatment and percutaneous coronary interventions for stable coronary heart disease, was not more effective than optimal medical therapy alone for preventing cardiovascular events, hospitalization or death, suggesting that drugs, surgical procedures or both were not a statistically effective solution for stable chronic angina. By inference, a therapeutic approach for mot severe coronary syndromes as UA, post- myocardial infarction angina, or aggravated angina episodes, seems to be a more distant goal.

Physiological Basis for Innovation: For more than a century, the extremely rapid coupled tissue O2/CO2 gas exchange and ion H/K transport by Hemoglobin (Hb) in red blood cell (RBC) has been well known for scientific community, the so-called Bohr/Haldane Effect (7). Since then, it has been noted and confirmed that RBC have a critical role to maintain normal vascular function, blood flow and tissue oxygenation and acid-base regulation. These functional roles of RBC include a nitric oxide (NO) transport, NO synthetasa, and regulation of platelet aggregation, vascular rheology, and endothelial function (8). Indeed, recent studies have demonstrated that erythrocyte serves as a regulator of vascular tone and tissue perfusion, whereas the hemoglobin and RBC itself may be sensors for the oxygen tissue requirement (9).

In this context, the evidence that erythrocytes are the major intravascular storage of nitrites (10), and that nitroglycerin effects on erythrocyte rheology and oxygen unloading in myocardial ischemia are mediated by S-Nitrosohemoglobin (11) implies that RBC K exchange should be preserved in subjects with CHD, especially if a hereditable defect in RBC K transport exists (12). Unfortunately, and despite such multiple integrated functions to maintain tissue oxygenation in health and diseases states, the role of RBC has never been considered in the therapeutic approach of stable chronic angina (13). However, our recent observation that reversal of an abnormal low RBC K content in hypertensive patients receiving low doses of pyrazinoylguanidine hydrochloride (amiloride HCl, 5 mg), and calcium gluconolactate was associated with a better control of BP, and regression of the ST-T alterations related to LVH or coronary heart disease (14), strongly support a novel mechanistic approaches to improve blood flow and myocardium oxygen transport in stable chronic angina.

Informed consent will be obtained in each patient, and the Review board committee of the Docent Institute of Urology, University of Carabobo Medical School, Valencia, will approve the trial. This trial is a continuation of the Protocol ID UIC-3 2007 (Novel Treatment for Coronary Artery Disease, NCT 01228214) and will be also registered in the ClinicalTrials.gov

METHODS

(I) Clinical Methods

At the inclusion period and in each clinical visit all subjects had measurements of BP, HR, body weight/height and measurement of body resistance and reactance for Body Composition Analysis of Total Body water and extra-cellular spaces, Fat-Free-Mass, Fat Mass. Number of anginal episodes, and functional anginal class (CCS) will be recorded in each case.

(II) Laboratory Methods

All patients will have routine measurement of Ion Transport Studies, which includes a 12-hour night (7 pm- 7 am) urine collection, followed by fasting state for measurement of plasma (Na, K, Cl, Mg++, Ionized calcium), RBC (Na, K, H2O content), and urine (Na, K, Cl, Mg++, calcium) electrolytes, along with plasma and urine osmolality, at entry, 4-week, and at 3, 8 and 12-months period.

(III) Cardiovascular Studies

All subjects All subjects had resting 12-lead ECG at entry, and non-invasive hemodynamic and PWA (DynaPulse200M, San Diego, CA) for Aortic Stiffness (Augmentation index, and Travel-Time-Reflected-Wave), Systemic and Brachial Artery Resistance and Compliances, obtained at entry and during clinical visits, including possible emergency attention. EchoC, or Doppler studies will be evaluated at baseline, 6-month, and 12-month periods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; age 35-75 years having angina (Canada Cardiovascular Society Class II-IV)
2. Essential Hypertension defined as taking at least 1 anti-hypertensive medication, or average systolic blood pressure ≥140 mm Hg, or diastolic blood pressure ≥90 mmHg
3. ST-T changes of LVH (Romhilt-Estes or Framingham Heart Study criteria, with typical LV strain pattern, or isoelectric, inverted or biphasic T waves)
4. ST-T changes of ischemia in resting ECG (ST depression, isoelectric, biphasic, negative or inverted T-waves)
5. Serum potassium < 5.0 mmol/L prior to randomization
6. Negative pregnancy test in child-bearing potential women
7. Willing to comply with scheduled visits
8. Informed consent form signed by the subject

Exclusion Criteria:

1. Resistance hypertension despite 3-drugs treatment
2. Myocardial infarction in past 90 days
3. Coronary artery bypass graft surgery in past 90 days
4. Atrial fibrillation with a resting heart rate > 90 bpm
5. Percutaneous coronary intervention in past 30 days
6. Implanted Pacemaker
7. Stroke in past 90 days
8. Left or Right Ventricular Branch Block
9. Aldosterone antagonist or K sparing drug in last 7 days
10. Intolerance to amiloride
11. Lithium use
12. Current participation in any other therapeutic trial
13. Any condition that may prevent the subject from adhering to the trial protocol
14. History of hyperkalemia (K ≥5.5 mmol/L) in the past six months or K >5.0 mmol/L within 2 weeks
15. Chronic renal dysfunction
16. Liver disease
17. Chronic pulmonary disease
18. Significant uncorrected valvular heart disease

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Regression of Angina without Recurrence | Baseline, and every 6-months therafter
  Evaluation of Angina Class according Canadian Cardiology Society (CCS)
Regression of ST-T and T-waves alterations of Myocardial Ischemia | Baseline and every 6-months thereafter
  Evaluation according Minnesota Code
RBC K Content | Baseline and very 6-Months thereafter
  Obtained by a novel accurate method developed in our laboratory (Nutr Metab Cardiovasc Dis. 2002 Jun;12(3):112-116

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Delgado-Leon, MD, Study Chair — University of Carabobo; Antonio R Delgado-Almeida, MD, FAHA, FACC, APS, Principal Investigator — Clinical Research Unit at Docent Institute of Urology; Carlos L Delgado-Leon, MD, Study Director — Venezuelan Foundation of Heart Failure
Locations (1):
- Hypertension Research Unit, Valencia, Carabobo, Venezuela

REFERENCES:
- [Background] ACC/AHA 2007 Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction. J Am Coll Cardiol, 2007; 50:1-157
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] Wald NJ, Law MR. A strategy to reduce cardiovascular disease by more than 80%. BMJ. 2003 Jun 28;326(7404):1419. doi: 10.1136/bmj.326.7404.1419. PMID 12829553
- [Background] Nicholls SJ, Tuzcu EM, Sipahi I, Grasso AW, Schoenhagen P, Hu T, Wolski K, Crowe T, Desai MY, Hazen SL, Kapadia SR, Nissen SE. Statins, high-density lipoprotein cholesterol, and regression of coronary atherosclerosis. JAMA. 2007 Feb 7;297(5):499-508. doi: 10.1001/jama.297.5.499. PMID 17284700
- [Background] Simons M, Annex BH, Laham RJ, Kleiman N, Henry T, Dauerman H, Udelson JE, Gervino EV, Pike M, Whitehouse MJ, Moon T, Chronos NA. Pharmacological treatment of coronary artery disease with recombinant fibroblast growth factor-2: double-blind, randomized, controlled clinical trial. Circulation. 2002 Feb 19;105(7):788-93. doi: 10.1161/hc0802.104407. PMID 11854116
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Jensen FB. Red blood cell pH, the Bohr effect, and other oxygenation-linked phenomena in blood O2 and CO2 transport. Acta Physiol Scand. 2004 Nov;182(3):215-27. doi: 10.1111/j.1365-201X.2004.01361.x. PMID 15491402
- [Background] Crawford JH, Isbell TS, Huang Z, Shiva S, Chacko BK, Schechter AN, Darley-Usmar VM, Kerby JD, Lang JD Jr, Kraus D, Ho C, Gladwin MT, Patel RP. Hypoxia, red blood cells, and nitrite regulate NO-dependent hypoxic vasodilation. Blood. 2006 Jan 15;107(2):566-74. doi: 10.1182/blood-2005-07-2668. Epub 2005 Sep 29. PMID 16195332
- [Background] Ellsworth ML, Forrester T, Ellis CG, Dietrich HH. The erythrocyte as a regulator of vascular tone. Am J Physiol. 1995 Dec;269(6 Pt 2):H2155-61. doi: 10.1152/ajpheart.1995.269.6.H2155. PMID 8594927
- [Background] Dejam A, Hunter CJ, Pelletier MM, Hsu LL, Machado RF, Shiva S, Power GG, Kelm M, Gladwin MT, Schechter AN. Erythrocytes are the major intravascular storage sites of nitrite in human blood. Blood. 2005 Jul 15;106(2):734-9. doi: 10.1182/blood-2005-02-0567. Epub 2005 Mar 17. PMID 15774613
- [Background] Bin JP, Doctor A, Lindner J, Hendersen EM, Le DE, Leong-Poi H, Fisher NG, Christiansen J, Kaul S. Effects of nitroglycerin on erythrocyte rheology and oxygen unloading: novel role of S-nitrosohemoglobin in relieving myocardial ischemia. Circulation. 2006 May 30;113(21):2502-8. doi: 10.1161/CIRCULATIONAHA.106.627091. Epub 2006 May 22. PMID 16717147
- [Background] Delgado-Almeida A, Delgado MC. Hereditability Defect in Red-Cell K in Hypertension. FASEB J. 2008; 22:968.8 (abstract). FASEB Experimental Biology 2008. April 5-9, San Diego, California
- [Background] Fuster V. The several faces of clinical trials: from new therapies to failed preventive strategies. Nat Clin Pract Cardiovasc Med. 2006 Apr;3(4):173. doi: 10.1038/ncpcardio0520. No abstract available. PMID 16568110
- [Background] Delgado-Almeida A, Delgado-Leon C, Delgado-Leon AJ. Amiloride and red blood cell potassium transport in coronary artery disease: Reversion of the clinical and ECG alterations (abstract). 2007 Scientific Meeting of the Inter-American Society of Hypertension and the Consortium for Southeastern Hypertension Control. Miami 6-10, 2007.
- [Background] Finimundi HC, Caramori PA, Parker JD. Effect of diuretic therapy on exercise capacity in patients with chronic angina and preserved left ventricular function. J Cardiovasc Pharmacol. 2007 May;49(5):275-9. doi: 10.1097/FJC.0b013e3180385ad7. PMID 17513945